CLINICAL TRIAL: NCT00384657
Title: The Effects of Intravenous Iron Therapy for Anemia Correction in Patients With Severe Chronic Heart Failure and Concomitant Moderate Chronic Kidney Disease
Brief Title: Intravenous Iron in Patients With Severe Chronic Heart Failure and Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of cooperation among centers, Financial reasons
Sponsor: Anemia Working Group Romania (Other)
Responsible Party: Principal Investigator, Liliana Garneata, Dr, Anemia Working Group Romania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWG_06_01
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Chronic Kidney Disease; Chronic Heart Failure; Anemia
Keywords: chronic heart failure; chronic kidney disease; anemia; intravenous iron
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): iv iron sucrose
  Interventions: Drug: iron sucrose
- Group II (No Intervention): Patients will receive conventional treatment of Chronic Heart Failure.

INTERVENTIONS:
Drug: iron sucrose — Patients in Group I will receive iv iron sucrose, as described in the study protocol.
  Patient in Group II will receive conventional treatment for chronic heart failure.
  Other Names: Group I - iv iron group; Group II - conventional treatment group
  Arms: Group I

SUMMARY:
Recently, growing body of evidence support the finding that anemia frequently occurs in patients with chronic heart failure (CHF). Chronic kidney disease (CKD), as well, is highly prevalent among heart failure patients, and both anemia and CKD are independently associated with increased mortality. A vicious circle is established with CHF causing both chronic renal insufficiency and anemia, and CKD further aggravating anemia which, in turn, worsens CHF and so on. Treatment of the anemia breaks this circle and improves the quality of life, cardiac and renal functions in patients with severe CHF.

Intravenous iron alone was proved to allow the maintenance of target hematocrit in one-third of chronic renal failure predialysis patients.

Based on these considerations, intravenous iron for anemia in patients with CHF and moderate CKD would represent a reasonable therapeutic approach.

The aim of the trial is to assess the efficiency of intravenous iron therapy in the management of mild to moderate anemia associated with CHF NYHA III class and concomitant moderate CKD.

DETAILED DESCRIPTION:
Intravenous iron administration in CHF patients with absolute or functional iron deficiency could correct their anemia, thus improving cardiac function judged by ejection fraction and NYHA functional class. If true, enhancement of cardiac output will increase oxygen delivery to tissues, including renal cortex. This might improve the renal functions and slow the rate of progression of CKD reflected by the slope of decline in glomerular filtration rate (GFR).

Since erythropoietin synthesis is located in peritubular fibroblasts from outer renal cortex, which is the most affected area during chronic hypoxia, increasing renal blood flow after anemia correction is expected to restore optimal erythropoietin production and normalize plasma Epo levels.

The primary objective is to assess the efficiency of intravenous iron therapy in the management of mild to moderate anemia associated with chronic heart failure NYHA III class and concomitant moderate chronic kidney disease.

The secondary objectives are to determine if the correction of anemia in these patients affects the cardiac function, the rate of progression of CKD and the plasma erythropoietin levels.

The study will be conducted in accordance with the Declaration from Helsinki and Tokyo, with the amendments from Venice (1983), after the approval by the local ethics committee.

The total observation period will be of 28 weeks, with a pre-study phase (selection, randomization of subjects) 4 weeks.The study period will last 24 weeks, with a possible extension to 48 weeks, depending on the results of this first phase.

200 anemic patients with chronic heart failure class NYHA III and concomitant stage 3 chronic kidney disease will be enrolled, after obtaining their written informed consent.

All patients will be evaluated for the inclusion and exclusion criteria at enrollment and at each visit during the pre-study phase. Only patients fulfilling all the requested criteria at all evaluation moments will be enrolled. The enrolled subjects will be centrally randomly assigned in a 1:1 ratio into two study groups.

Group I (treatment group): Subjects assigned to this group will receive intravenous iron (ferric sucrose product Venofer® 2%, 5mL/ampoule) in a starting dose of 200mg (2 ampoules) diluted in 150mL 0.9% NaCl solution, over 60 minutes, once a week for the first four administrations, and then every other week until hemoglobin levels reach 12g/dL. Then, iron dose will be adjusted to 1 ampoule at 2-4 weeks interval, as needed to maintain these levels with serum ferritin ≤500ng/mL.

Iron administration will be discontinued if serum ferritin will exceed 500ng/mL, and will be restarted with a reduced dosage (1 ampoule at every 2-4 weeks) once serum ferritin decrease below this value.

Conventional treatment for CHF will be continued as needed. Group II (control group): Subjects assigned to this group will continue their conventional treatment for CHF as needed, without iron supplementation.

No other anti-anemic medication will be administered in either group during the study period.

Subject's visits will take place at two weeks intervals in the first 12 weeks of the study phase and at 4 weeks apart thereafter. At each visit will be recorded, according to the schedule, data concerning physical examination, including signs of CHF, hematological and iron status, renal function, concomitant medication and adverse events.

Parameters recorded at the time of first iron administration will serve as baseline determination.

The completion of the study will be declared when 200 subjects will complete the whole observation period, according to the above protocol.

ELIGIBILITY:
Inclusion Criteria:

* persistent severe CHF: functional class NYHA III (marked limitation of physical activity - comfortable at rest, but less than ordinary activity results in shortness of breath and/or fatigue16); left ventricular ejection fraction (echocardiography) less than 40%; functional and systolic dysfunction criteria must be stable at two different examinations one month apart;
* stable stage 3 chronic kidney disease: estimated GFR between 30-59mL/min/1.73m2 (mean value of three measurements within the last 8 weeks, separated from each other by at least one week); stable renal function (at least three different measurements within the past 8 weeks, separated from each other by at least one week; the difference between the highest and the lowest value should be less than 5mL/min/1.73m2)
* mild to moderate anemia: hemoglobin levels < 12g/dL (mean value of three measurements within the last 8 weeks, separated from each other by at least one week) and stable (at least three measurements within the last 8 weeks; the difference between the highest and the lowest value should be less than 1.5g/dL);
* iron deficiency: absolute (serum ferritin < 100ng/mL) or functional (serum ferritin 100-300ng/mL and transferrin saturation < 20%)

Exclusion Criteria:

* evidence of active gastrointestinal or genital tract bleeding
* folate or vitamin B12 deficiency
* hypothyroidism
* hemolytic anemia
* any primary kidney diseases (glomerulonephritis, interstitial nephritis, cystic diseases)
* systemic diseases with renal involvement (lupus erythematosus, vasculitis, amyloidosis)
* renal artery stenosis (>70% lumen reduction)
* diabetic nephropathy
* severe malnutrition (SGA score C or lower)
* active liver diseases
* infectious conditions
* malignancies
* C-reactive protein > 12 mg/L
* severe anemia (< 8.5g/dL)
* blood transfusions in the preceding two months
* iron therapy in the preceding three months
* concomitant erythropoietin therapy
* severe arterial hypertension (systolic BP >190 mm Hg and/or diastolic BP >115 mm Hg)
* recent history (less than 3 months) of acute coronary syndrome
* recent (less than 1 month) PCI
* recent (less than 1 month) CABG surgery
* active myocarditis
* active endocarditis
* more than mild valvar stenosis
* more than moderate valvar (mitral or aortic) regurgitation
* uncontrolled haemodynamically relevant atrial fibrillation/flutter
* hypertrophic cardiomyopathy
* acute and/or chronic pericarditis
* cor pulmonale
* participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
percentage of patients with increased ejection fraction | 12 months

SECONDARY OUTCOMES:
the need for blood transfusions during the study period | 12 months
serum ferritin level | 12 months
transferrin saturation | 12 months
radial myocardial velocities | 12 months
right ventricular function | 12 months
global diastolic function | 12 months
left ventricular mass index | 12 months
major cardiovascular events (myocardial infarction, acute pulmonary edema, stroke) | 12 months
hospital admissions | 12 months
death of the patient (all causes deaths, cardiac deaths) | 12 months
slope of GFR change | 12 months
"death" of the kidney (initiation of renal replacement therapy) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Professor, Study Director — Dr Carol Davila Teaching Hospital of Nephrology; Tiberiu Nanea, Professor, Principal Investigator — "Caritas" Teaching Hospital, Bucharest; Liliana Garneata, MD, PhD, Principal Investigator — Dr Carol Davila Teaching Hospital of Nephrology Bucharest
Locations (2):
- Romania (2):
  - "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest
  - "Caritas" Teaching Hospital, Cardiology Department, Bucharest